CLINICAL TRIAL: NCT03976583
Title: Remineralization Potential of Pearl Powder Compared to CPP-ACP on Enamel White Spot Lesions (Randomized Controlled Trial)
Brief Title: Remineralization Potential of Pearl Powder Compared to CPP-ACP on Enamel White Spot Lesions
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shereen Assem El-Sherif, Assistant Lecturer - Conservative Department- Faculty of Dentistry - MSA University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1081988
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: White Spot Lesion
MeSH Terms: interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex; pearl powder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cpp-acp (Active Comparator): MI paste Self-administration of the product by the patient once in the evening. A pea-size amount of the product should be applied per arch, using a dry finger or cotton pellet to distribute it evenly across all teeth and to work it into the interdental spaces. The product was then retained in the mouth for 1-3 min, and manipulated around the teeth using the tongue, before being expectorated and patient should not rinse it until 30 min.
  Interventions: Drug: Cpp-Acp
- Pearl powder (Experimental): Pure pearl powder in the form of gel Self-administration of the product should be used once daily (in the evening), after a 2 min manual tooth brushing. .Participants were explicitly instructed to apply the gel by his finger allover the teeth and not to rinse their mouths after application and not to eat or drink for at least 30 min.
  Interventions: Other: Pearl powder

INTERVENTIONS:
Drug: Cpp-Acp — Remineralising agent
  Other Names: MI paste
  Arms: Cpp-acp
Other: Pearl powder — Natural product
  Arms: Pearl powder

SUMMARY:
The aim of this study is to evaluate the remineralization potential of pearl powder on early ('white spot') lesions in enamel in orthodontic patients compared to casein phosphopeptide-amorphous calcium phosphate.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the remineralization potential of pearl powder on early ('white spot') lesions in enamel in orthodontic patients compared to casein phosphopeptide-amorphous calcium phosphate. The remineralisation potential will be assessed both visually and by standardised photographic image analysis. the follow up will be up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Males or females.
* Age: 12-25 years old.
* Patients with good oral hygiene.
* Co-operative patients who show interest to participate in the study.

Exclusion Criteria:

* Patients with bad oral hygiene.
* Lack of patient's approval and compliance.
* Presence of abnormal oral, medical, or mental condition.
* Patients who are allergic to milk products.
* Pregnant and lactating women.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical index used for visual evaluation of white spot lesions | 12 months
  Scores(0-No visible colour change, 1-Slight white colour change, only visible after air-drying, 2-Slight colour change with certain marked white areas, 3-White consistent colour change, 4-Distinct white colour change)

SECONDARY OUTCOMES:
Digital photographic image analysis | 12 months
  Computerised software to analyse the change in the lesion